CLINICAL TRIAL: NCT02612298
Title: Efficacy and Safety of Arotinolol Hydrochloride on Morning Blood Pressure and Heart Rate in Patients With Essential Hypertension
Brief Title: Efficacy and Safety of Arotinolol Hydrochloride on Morning Blood Pressure and Heart Rate
Acronym: ESAHOM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sumitomo Pharma (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSPC-ALM-1401
Record Dates: First submitted 2015-09-02; First posted 2015-11-23 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Essential Hypertension
Keywords: Essential Hypertension; Arotinolol; Morning Blood Pressure
MeSH Terms: conditions — Essential Hypertension | interventions — arotinolol; Almarl; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- arotinolol (Experimental): Arotinolol Hydrochloride, oral, 5-15mg, bid for 12 weeks
  Interventions: Drug: Arotinolol Hydrochloride
- Metoprolol (Active Comparator): Metoprolol succinate sustained-release tablet, oral, 23.75-71.25mg, qd for 12 weeks.
  Interventions: Drug: Metoprolol succinate sustained-release tablet

INTERVENTIONS:
Drug: Arotinolol Hydrochloride — Arotinolol Hydrochloride, oral, 5-15mg, bid for 12 weeks.
  Other Names: Almarl
  Arms: arotinolol
Drug: Metoprolol succinate sustained-release tablet — Metoprolol succinate sustained-release tablet,oral, 23.75-71.25mg, qd for 12 weeks.
  Other Names: Betaloc tablet
  Arms: Metoprolol

SUMMARY:
The purpose of this study is to compare the efficacy and safety of Arotinolol Hydrochloride and Metoprolol succinate on morning blood pressure, heart rate and target organ damage in patients with essential hypertension. To provide evidence for hypertension treatment.

A group: Arotinolol Hydrochloride, oral, 5-15mg, bid for 12 weeks. B group: Metoprolol succinate sustained-release tablet, oral, 23.75-71.25mg, qd for 12 weeks.

DETAILED DESCRIPTION:
Compare the efficacy and safety of Arotinolol Hydrochloride and Metoprolol succinate on morning blood pressure, heart rate and target organ damage in patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with systolic blood pressure between 140-179mmHg and/or diastolic blood pressure between 90-109mmHg.
2. Aged between 18-65 years old.
3. Signed informed consent.

Exclusion Criteria:

1. Secondary hypertension
2. Patients who taking amiodarone over 200mg/day to control arrhythmia
3. Patients who taking class I antiarrhythmic drugs
4. Resting heart rate less than 60bpm
5. Serious liver and kidney disease: aspartate aminotransferase (AST) or alanine aminotransferase) (ALT)>2.5 times upper limit of normal; serum creatinine>3mg/dl (265umol/L)
6. Severe heart failure: New York Heart Association (NYHA) functional class 2, 3, 4
7. Myocardial infarction or stroke in the last three months. Unstable angina pectoris in the last month.
8. Patients with asthma or chronic obstructive pulmonary disease.
9. Pregnancy and breast-feeding
10. Patients allergy to investigational drugs or have contraindication to investigational drugs.
11. Others unsuitable to participate in the study judged by investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

PRIMARY OUTCOMES:
Diastolic blood pressure | 12 weeks
  Changes in diastolic blood pressure measured by ambulatory blood pressure monitoring (ABPM) after treatment

SECONDARY OUTCOMES:
Systolic blood pressure | 12 weeks
  Changes in systolic blood pressure measured by ABPM after 12 weeks of treatment
Morning surge | 12 weeks
  Changes in morning surge after 12 weeks of treatment
The increase rate of morning blood pressure | 12 weeks
  Changes in the increase rate of morning blood pressure after 12 weeks of treatment
Morning blood pressure (BP) by office BP measure | 12 weeks
  Changes in morning blood pressure by office BP measure after 12 weeks of treatment
Heart rate by office BP measure | 12 weeks
  Changes in heart rate by office BP measure after 12 weeks of treatment
Pulse wave velocity (PWV) | 12 weeks
  Changes in PWV after 12 weeks of treatment
Ankle-brachial index (ABI) | 12 weeks
  Changes in ABI after 12 weeks of treatment
Albumin-to-creatinine ratio (ACR) | 12 weeks
  Changes in ACR after 12 weeks of treatment
Glomerular filtration rate (GFR) | 12 weeks
  Changes in GFR after 12 weeks of treatment

OTHER OUTCOMES:
Safety assessed by incidence rate of adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- China PLA General Hospital, Beijing, China